CLINICAL TRIAL: NCT00452439
Title: A Randomized, Double Blinded Study of Actonel for the Prevention of Bone Loss in Patients Receiving High Dose Corticosteroids for the Treatment of Acute Lymphocytic Leukemia (ALL) and Lymphoblastic Lymphoma (LL)
Brief Title: A Study of Actonel for the Prevention of Bone Loss
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0124; NCI-2010-01997 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Leukemia; Lymphoma
Keywords: Leukemia; Lymphoma; Acute Lymphocytic Leukemia; Lymphoblastic Lymphoma; Actonel; Risedronate; Bone Loss; Osteoporosis
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Bone Diseases, Metabolic; Osteoporosis | interventions — Risedronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actonel (Active Comparator): Actonel (Risedronate) + Vitamin D + Calcium
  Interventions: Drug: Actonel (Risedronate); Dietary Supplement: Calcium; Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo + Vitamin D + Calcium
  Interventions: Dietary Supplement: Calcium; Dietary Supplement: Vitamin D

INTERVENTIONS:
Drug: Actonel (Risedronate) — 35 mg (pill) by mouth weekly
  Other Names: Risedronate Sodium
  Arms: Actonel
Dietary Supplement: Calcium — 500 mg by mouth twice a day for a total of 24 months.
Dietary Supplement: Vitamin D — 400 IU by mouth twice a day for a total of 24 months.

SUMMARY:
The goal of this clinical research study is to learn if Actonel (risedronate) can help to prevent the development of osteoporosis (brittle and weak bones) caused by the steroid medication used to treat leukemia. The safety of this treatment in patients with ALL or LL will also be studied.

DETAILED DESCRIPTION:
One of the side effects of using high dose corticosteroids for the treatment of ALL is osteoporosis. Risedronate is a medication that was designed to help prevent osteoporosis (brittle and weak bones).

Before treatment you will receive a complete physical exam. You will have around 1 tablespoon of blood drawn for blood tests (these tests are in addition to the routine blood tests you will have as part of the treatment for leukemia). You will have a urine sample collected for routine tests. You will also have a bone mineral density test. This test measures the density of the bones in your spine, hip, and total body. The test is similar to having x-rays of your bones taken.

You will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in the first group will be given risedronate (once per week), vitamin D (once per day), and calcium (once per day). All three medications are pills and will be taken by mouth. Participants in the second group will be given placebo (once per week), vitamin D (once per day), and calcium (once per day). All three medications are pills and will be taken by mouth. A placebo is a substance that looks like the study drug but has no active ingredients. Neither you nor your doctor will know to which group you are assigned. However, if it is needed for your care, the information will be given to your doctor.

Participants in both groups will continue to receive chemotherapy during this study as scheduled. During chemotherapy, you will have around 1 tablespoon of blood drawn every 1-2 weeks for routine blood tests (as part of the standard of care for your treatment of leukemia).

For this study, you will have urine samples collected and repeat bone mineral density tests 6 months, 12 months, 18 months, and 24 months after starting the study drug (or placebo).

If you develop intolerable side effects from the risedronate you will be taken off the study.

This is an investigational study. Risedronate is FDA approved and commercially available. Up to 80 eligible patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Newly diagnosed ALL or LL receiving chemotherapy with augmented BFM, Hyper-CVAD or any variant of hyper-CVAD.
3. Female patients of childbearing potential (i.e. no hysterectomy, no loss of menses for 12 consecutive months), must be willing to use contraception.
4. Negative pregnancy test in female patients.
5. Patients must be enrolled within 6 weeks of starting induction chemotherapy.

Exclusion Criteria:

1. Hypocalcemia of less than 8.4 (corrected to account for the albumin level, [see Appendix E for formula])
2. Hypersensitivity to risedronate or other bisphosphonates
3. Inability to sit or stand upright for at least 30 minutes
4. Bone density T-score of -2.5 S.D or less.
5. Renal insufficiency (calculated creatinine clearance <30cc/min,[see Appendix F for formula])
6. Patients with a 25-hydroxyvitamin D concentration of less than 20 ng/ml and evidence of osteomalacia (low ionized calcium and high intact PTH).
7. Concomitant use of bisphosphonates, calcitonin, anabolic steroids, or fluoride.
8. Corrected calcium above 10.2, due to a cause not related to leukemia/lymphoma (i.e. hyperparathyroidism, multiple myeloma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2004-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria E. Cabanillas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: February 06, 2004 to March 10, 2010. All participants were recruited at University of Texas (UT) MD Anderson Cancer Center.
Groups:
- Actonel: Actonel (Risedronate) + Vitamin D + Calcium
  Actonel 35 mg orally weekly, Calcium 500 mg orally twice a day, and Vitamin D 400 IU orally twice a day for a total of 24 months.
- Placebo: Placebo + Vitamin D + Calcium
  Placebo weekly, Calcium 500 mg orally twice a day, and Vitamin D 400 IU orally twice a day for a total of 24 months.
Period: Overall Study
Arm/Group | Actonel | Placebo
Started | 36 | 36
Completed | 22 | 29
Not Completed | 14 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Refused Treatment | 4 | 3
Not completed — Death | 3 | 1
Not completed — Bone Marrow Transplant | 0 | 1
Not completed — Too Ill to Continue | 0 | 1
Not completed — Failed to achieve complete response | 2 | 0
Not completed — Relapse | 3 | 0
Not completed — Fracture | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Actonel | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Median (Full Range); unit: years] | 29 [23 to 49] | 42 [26 to 53] | 36 [23 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 24 | 21 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 17 | 35
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 36 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Bone Loss Reduction: Mean Percent Changes in BMD for Each Treatment Arm at the 6 Months
Description: bone mineral density (BMD) Mean percent Change in Bone Density from Baseline to 6 months.
Time Frame: 6 months
Population: Of 72 randomized, 22 participants in risedronate & 29 in placebo had at least a 6-month follow-up bone mineral density and were considered evaluable for the primary endpoint. Only 12/22 patients (55%) in risedronate and 7/29 patients (24%) in the placebo arm had 12 month DXA scan performed, mostly due to significant decreases in bone density.
Measure: Mean (Standard Deviation); unit: Percent of change
Arm/Group | Actonel | Placebo
Number analyzed (Participants) | 22 | 29
Percent of change
  Lumbar Spine 6 Months | -2.4 (0.05) | -3.5 (0.04)
  Right Hip 6 Months | -7.6 (0.06) | -11 (0.06)
  Left Hip 6 Months | -8.2 (0.06) | -11 (0.06)

2. Primary Outcome: Bone Loss Reduction: Mean Percent Changes in BMD for Each Treatment Arm at 12 Months
Description: bone mineral density (BMD) Mean percent Change in Bone Density from Baseline to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Actonel | Placebo
Number analyzed (Participants) | 12 | 7
percentage of change
  Lumbar Spine 12 Months | -0.6 (0.05) | -5 (0.05)
  Right Hip 12 Months | -4.8 (0.05) | -5.8 (0.05)
  Left Hip 12 Months | -4.1 (0.05) | -7 (0.03)

ADVERSE EVENTS:
Time Frame: Up to 6 years
Arm/Group | Actonel | Placebo
All-Cause Mortality (participants affected / at risk) | 3/36 | 1/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes